CLINICAL TRIAL: NCT02054546
Title: Novel Biomarkers (TIMP-2 and IGFBP7) of Tubular Renal Cell Damage for the Prediction of the Cardiac Surgery Associated Acute Kidney Injury (CSA-AKI) - A Feasibility Study
Brief Title: TIMP-2 and IGFBP7 for the Prediction of the Cardiac Surgery Associated Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 514/13
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to analyze the new biomarkers (TIMP-2 and IGFBP-7) of tubular renal cell damage for the prediction of the Cardiac Surgery Associated acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* planned cardiac surgery

Exclusion Criteria:

* renal dialysis
* minors
* emergency
* no cardiopulmonary bypass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with planned cardiac surgery and cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
AKI-stadium 1 (KDIGO) | 30 days

SECONDARY OUTCOMES:
all cause mortality | 30 days

OTHER OUTCOMES:
AKI Stadium 2-3 (KDIGO) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jens Fassl, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Universitätsspital Basel, Basel, Canton of Basel-City, Switzerland